CLINICAL TRIAL: NCT06273930
Title: Reduction of Dentine Hypersensitivity After Non-surgical Periodontal Therapy Comparing 5% Calcium Sodium Phosphosilicate and 8% Arginine Dentifrices: a Single Centre, Randomized Control Trial
Brief Title: Reduction of Dentine Hypersensitivity After Use of Different Dentifrices
Acronym: Dentrifices
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Muhammad Junaid Iqbal, Principle investigator, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AFID
Record Dates: First submitted 2024-02-05; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Sensitivity, Tooth
MeSH Terms: conditions — Dentin Sensitivity | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): Superiority parallel 3-arm randomized control trial. The intention behind a superiority trial is that CSPS & Arginine are superior to commercially available desensitizing agents.
  Double blinded study (Participants and Outcome Assessor)
  Allocation ratio 1:1:1
  Patients are chosen based on inclusion criteria. Patients undergo non-surgical periodontal therapy as part of their treatment. DH is assessed using the Schiff scale evaluation and tactile test Visual analogue Score (VAS) after treatment.
  2 groups of patients receiving desensitizing agents applied for two consecutive 3-second applications, while others are placed in a control group.
  DH is evaluated again immediately using the Schiff scale and tactile test VAS after the application of desensitizing agents Patients are instructed to maintain their oral hygiene by brushing their teeth twice daily with a specific dentifrice provided to them along with a soft toothbrush.
- 5% CSPS group (Active Comparator): Superiority parallel 3-arm randomized control trial. The intention behind a superiority trial is that CSPS & Arginine are superior to commercially available desensitizing agents.
  Double blinded study (Participants and Outcome Assessor)
  Allocation ratio 1:1:1
  Patients are chosen based on inclusion criteria. Patients undergo non-surgical periodontal therapy as part of their treatment. DH is assessed using the Schiff scale evaluation and tactile test Visual analogue Score (VAS) after treatment.
  2 groups of patients receiving desensitizing agents applied for two consecutive 3-second applications, while others are placed in a control group.
  DH is evaluated again immediately using the Schiff scale and tactile test VAS after the application of desensitizing agents Patients are instructed to maintain their oral hygiene by brushing their teeth twice daily with a specific dentifrice provided to them along with a soft toothbrush.
  Interventions: Drug: 5% CALCIUM SODIUM PHOSPHOSILICATE
- 8% arginine group (Active Comparator): Superiority parallel 3-arm randomized control trial. The intention behind a superiority trial is that CSPS & Arginine are superior to commercially available desensitizing agents.
  Double blinded study (Participants and Outcome Assessor)
  Allocation ratio 1:1:1
  Patients are chosen based on inclusion criteria. Patients undergo non-surgical periodontal therapy as part of their treatment. DH is assessed using the Schiff scale evaluation and tactile test Visual analogue Score (VAS) after treatment.
  2 groups of patients receiving desensitizing agents applied for two consecutive 3-second applications, while others are placed in a control group.
  DH is evaluated again immediately using the Schiff scale and tactile test VAS after the application of desensitizing agents Patients are instructed to maintain their oral hygiene by brushing their teeth twice daily with a specific dentifrice provided to them along with a soft toothbrush.
  Interventions: Drug: 8% Arginine

INTERVENTIONS:
Drug: 5% CALCIUM SODIUM PHOSPHOSILICATE — Calcium sodium phosphosilicate is a particulate, bioactive glass material that degrades in the aqueous oral environment to release calcium and phosphate ions, leading to formation of hydroxycarbonate apatite on the dentine surface result in reduction in dentine hypersenstivity
  Arms: 5% CSPS group
Drug: 8% Arginine — Arginine contributes to Whole Mouth Health. It also plays a role with respect to dental caries, helping to maintain a pH-neutral environment, and is proven to rapidly help relieve dentin sensitivity. Arginine is truly a remarkable ingredient now being used in oral care products.
  Arms: 8% arginine group

SUMMARY:
To assess the impact of the use of 5% Calcium Sodium Phosphosilicate or 8% Arginine dentifrices on dentinal hypersensitivity following non-surgical periodontal therapy in patients with periodontitis.

DETAILED DESCRIPTION:
To assess the impact of the use of 5% Calcium Sodium Phosphosilicate or 8% Arginine dentifrices on dentinal hypersensitivity following non-surgical periodontal therapy in patients with periodontitis. patients will be selected on the bases of inclusion and exclusion criteria.Descriptive statistics will be presented for both qualitative and quantitative variables

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be between 30 and 65 years old.
2. Participants should be in good general health.
3. Participants must have a diagnosis of generalized chronic periodontitis according to the 1999 classification definition.
4. Participants should complain of at least two teeth with dentinal hypersensitivity.
5. Participants must exhibit moderate to severe dentinal hypersensitivity (Schiff's scores of 2 to 3) or tactile stimulation (Visual Analogue Scale (VAS) score >4) after at least one scaling and root planing session.

Exclusion Criteria:

1. Individuals with dentinal hypersensitivity symptoms prior to periodontal treatment.
2. Those who have used agents to treat hypersensitivity in the past 3 months.
3. Participants who are allergic to the test products (5% CSPS or 8% arginine).
4. Dentinal hypersensitivity caused by factors such as dental caries, defective restorations, fractured teeth, abrasion or abfraction, extensively restored teeth, or restorations extending into the test area.
5. Individuals who have undergone orthodontic treatment within the past 3 months.
6. Patients with crowded teeth or serving as abutment teeth for fixed or removable prostheses are also excluded from the study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
To assess the impact on Dentinal hypersensitivity following the use of 5% CSPS or 8% Arginine following non-surgical periodontal therapy in patients with Periodontitis by VAS. | within 8 weeks from the start of procedure
  Define pain and discomfort via running a probe on dentine of tooth The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health) orientated from the left (worst) to the right (best). In some studies, horizontal scales are orientated from right to left.
To assess the impact on Dentinal hypersensitivity following the use of 5% CSPS or 8% Arginine following non-surgical periodontal therapy in patients with Periodontitis by Schiff scale. | within 8 weeks from the start of procedure
  Schiff Cold Air Sensitivity Scale: is a tool used to assess dentinal hypersensitivity (DH) or tooth sensitivity to cold air. It's a clinical method developed to quantify the severity of cold air sensitivity experienced by individuals with dentin hypersensitivity.
  The scale typically ranges from 0 to 3, with the following descriptions:
  0: No response to cold air
  1. Mild, brief, or localized response to cold air
  2. Moderate response to cold air, patient can tolerate
  3. Severe and prolonged response to cold air, patient finds it intolerable

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad J Iqbal, Principal Investigator — AFID
Locations (1):
- AFID, Rawalpindi, Pakistan